CLINICAL TRIAL: NCT06097520
Title: Virtual Reality in Postoperative Acute Pain Management in Thoracic Surgery (VRThx)
Brief Title: Virtual Reality in Postoperative Acute Pain Management in Thoracic Surgery
Acronym: VRThx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-01673; am23Eckstein
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
Keywords: thoracic surgery; Virtual reality (VR)
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: investigator-initiated, single-center, randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Patients receive a VR headset (Pico G2 4K) for 15 minutes in the time between the 2. and 3. pain assessment and will experience non-interactive videos with different immersive scenarios of nature scenes. Nature sounds, meditation or classical music accompanying the scenarios are played through noise-cancelling headphones. Additionally, a wearable with an optical PPG- and EDA-Sensor (Empatica EmbracePlus) is put on the wrist of each participant in both groups 15 minutes before the inhalation until 15 minutes after the third pain intensity assessment, which enables the tracking of vital signs and monitoring of physiological responses. In both groups the study procedure starts with determining the pain intensity immediately before and after the 15 minutes inhalation procedure which is part of the standard of care. 15 minutes after the second assessment, the pain intensity is determined a third time in both groups.
  Interventions: Other: VR Intervention
- Control group (standard care) (No Intervention): Patients in the control group do not receive any intervention in the time between the second and third pain assessment. Additionally, a wearable with an optical PPG- and EDA-Sensor (Empatica EmbracePlus) is put on the wrist of each participant in both groups 15 minutes before the inhalation until 15 minutes after the third pain intensity assessment, which enables the tracking of vital signs and monitoring of physiological responses. In both groups the study procedure starts with determining the pain intensity using the Numeric Rating Scale (NRS) immediately before and after the 15 minutes inhalation procedure which is part of the standard of care. 15 minutes after the second assessment, the pain intensity is determined a third time in both groups.

INTERVENTIONS:
Other: VR Intervention — For the VR Intervention a VR head-mounted display, the Pico G2 4K, will be used. This intervention involves wearing VR glasses and experiencing non-interactive videos with sound through a headset. The footage consists of different immersive 360-degree scenarios from natural environments (e.g., forest), while corresponding sounds, meditation or classical music harmoniously tuned to these scenarios and are played through noise-cancelling headphones.
  Arms: Intervention group

SUMMARY:
This randomized controlled study is to investigate the effectiveness of VR headsets in reducing postoperative pain intensity among patients after having undergone thoracic surgical procedures.

DETAILED DESCRIPTION:
Thoracic surgical procedures can often result in postoperative pain. Traditional methods of pain management, such as medication, have limitations in terms of their efficacy and potential side effects. Therefore, there is a need for alternative approaches that can effectively alleviate postoperative pain while minimizing medication use. Virtual reality (VR) technology has gained attention as a potential non-pharmacological intervention for pain management. There is limited research specifically focusing on the use of VR in the context of thoracic surgery. This study is to investigate the effectiveness of VR headsets in reducing postoperative pain intensity among patients after having undergone thoracic surgical procedures. To enhance the objectivity of the investigation, objective parameters alongside subjective assessments of pain will be incorporated. While self-reported measures are valuable, they can be subjective and influenced by individual perception. Therefore, the subjective assessments will be complemented by objective measurements to gain a more comprehensive understanding of the pain experience and its modulation through the VR intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Written informed consent as documented by signature from the patient
* Video-assisted anatomical resection of the lung (VATS) (Surgery duration of at least 90 minutes)
* Ability to speak, understand and read German

Exclusion Criteria:

* Significant mental, cognitive or neurological impairments (Delirium, psychoses, unstable dissociative disorders, any form of organic brain disorder, …)
* Inability to follow the study procedures (e.g., due to language problems, visual and hearing impairments)
* Chronic pain
* Morphine intolerance
* Excessive alcohol consumption (men > 3 standard drinks, women > 2 standard drinks per day)
* Substance abuse
* Unable or not willing to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain intensity level | At first, second and third postoperative day: before the inhalation procedure, immediately after the inhalation and 15 minutes after the inhalation procedure
  Pain intensity will be measured using the Numeric Rating Scale (NRS). The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable".

SECONDARY OUTCOMES:
Opioid Consumption | 3 postoperative days
  Opioid consumption will be documented in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Timiliotis, MSc, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland